CLINICAL TRIAL: NCT00958477
Title: Phase I, Open-label Study to Investigate Safety, Tolerability, PK, and PD of EMD 525797 After Single and Repeated Dosing at Different Dose Levels in Subjects With Hormone-resistant Prostate Cancer With Bone Mets and Progressive Disease Following Prior CTX
Brief Title: A Study to Determine the Safety, Tolerability, Pharmacokinetics and Dynamic Effects of Different Doses of the Study Drug EMD 525797 in Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMR62242_002
Record Dates: First submitted 2009-08-11; First posted 2009-08-13 (Estimated); Results first posted 2017-08-02 (Actual); Last update posted 2017-08-02 (Actual); Status verified 2017-03

CONDITIONS: Prostate Cancer; Bone Metastases
Keywords: Safety; tolerability; pharmacokinetics; pharmacodynamics of EMD 525797; prostate cancer patients
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abituzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EMD 525797 (Experimental)
  Interventions: Biological: EMD 525797

INTERVENTIONS:
Biological: EMD 525797 — Subjects will be administered with 250 milligram (mg), 500 mg, 1000 mg or 1500 mg of EMD 525797 intravenously over 1 hour every 2 weeks for 6 weeks. Subjects who will be clinically benefitted at the end of week 6 were continued at the same dose-level until disease progression, intolerance to treatment, withdrawal of consent or if the subject is no longer benefitted from the treatment as per Investigator's discretion.

SUMMARY:
This study is intended to test an experimental new drug called, EMD 525797 (Study Drug). This drug is not yet approved for sale and has only been tested in a small number of people to date (prior to this study starting another research study was carried out involving 37 healthy volunteers receiving the Study Drug). Until more is known about this Study Drug, it can only be used in research studies.

This research study is planned to answer important questions about how the Study Drug is tolerated and how it may work in patients with prostate cancer with bone metastases.

This is a small study which is expected to include 24 patients, and will be conducted in approximately 3 hospitals in Germany and 1 hospital in Brussels, Belgium. The study will last until the last patient has had their last study visit which is expected to be about 18 months in total.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed written informed consent
* Age superior or equal to 18 years
* Subjects with histological or cytologically proven prostate cancer with evidence of bone metastases on bone scans or CT / MRI after prior chemotherapy with e.g. taxane or mitoxantrone Patients should have undergone bilateral orchiectomy or should be on continuous androgen deprivation therapy with a gonadotropin releasing hormone agonist or antagonist and should have stopped any anti-androgen therapy for at least 4 weeks before inclusion in the study. Patients should be either on stable (i.e., since at least 3 months) ongoing therapy with a bisphosphonate or without any bisphosphonate therapy. Initiation of a bisphosphonate therapy within this time period prior the study or during the study is not allowed. Total serum testosterone should be less than 50 ng/dL or 1.7 nmol/L.
* Evidence of progressive disease, defined by at least two PSA values above the individual nadir level with an increase of at least 10% each determined at a minimum interval of 2 weeks before screening examination. Presence of a measurable lesion is not required for study entry. Nodal (in lymph nodes superior or equal to 2cm) or visceral progression is sufficient for trial entry independent of PSA.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2 at study entry and an estimated life expectancy of at least 3 months.
* Adequate hematological function, defined by white blood cell count (WBC) greater than or equal to 3 x 109/L with absolute neutrophil count (ANC) greater than or equal to 1.5 x 109/L, and lymphocyte count greater than or equal to 0.5 x 109/L; platelet count greater than or equal to 100 x 109/L; and hemoglobin greater than or equal to 9 g/dL.
* Adequate hepatic function defined by total bilirubin level less than or equal to 1.5 times the upper limit of normal (ULN), and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels less than or equal to 2.5 x ULN; or, for subjects with documented metastatic disease to the liver, AST and ALT levels less than or equal to 5 x ULN.
* Adequate renal function defined by serum creatinine less than 1.5 mg/dL.
* Effective contraception. If the risk of conception exists, pregnancy has to be avoided during the study (SCR to EOS) as well as during at least 3 month after last dosing using an effective contraception method (e.g. double barrier method)

Exclusion Criteria:

* Any systemic cytotoxic cancer treatment within 4 weeks before treatment with EMD 525797.
* Acute pathologic fracture, spinal cord progression, hypercalcemia (within 4 weeks period prior to screening).
* Radiotherapy to bone lesions, orthopaedic surgery, or any investigational drug in the 30 days before the start of treatment in this study and during treatment period, and/or biopsies involving bone within 2 weeks before the start of treatment in this study.
* Supraphysiologic doses of steroids (defined as superior or equal to 7.5 mg of prednisone equivalents per day).
* Previous treatment with anti-integrin therapy.
* Confirmed or clinically suspected brain metastases.
* Known hypersensitivity reactions to any of the components of the study medication.
* History of allergic reactions to other monoclonal antibody (mAb) therapy.
* Uncontrolled hypertension (systolic greater or equal to 160 mmHg, diastolic greater than or equal to 100 mmHg).
* Current history of chronic daily aspirin therapy (ASS at doses inferior or equal to 100 mg is permitted), bleeding disorders and/or history of thromboembolic events (history of superficial thrombophlebitis is not an exclusion criterion); thrombolytics or oral or parenteral anticoagulants within 10 days prior to study start and during treatment period.
* Severe peripheral vascular disease or ulceration.
* Unstable angina pectoris, or myocardial infarction within 6 months before start of study treatment, clinical significant abnormal ECG at screening
* Known alcohol or drug abuse.
* Participation in another clinical trial within the past 30 days before start of study treatment.
* Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent.
* Ongoing uncontrolled infections, including active or chronic hepatitis B or C, ongoing HIV infection.
* Legal incapacity or limited legal capacity.
* All other significant diseases which, in the opinion of the Investigator, might impair the subject's tolerance of study treatment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2008-10; Primary Completion 2010-09 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Uhl, Dr, Dipl. Chem., Physician, Study Director — Merck KGaA, Darmstadt, Germany
Locations (4):
- Institut Jules Bordet - Medical Oncology Clinic, Brussels, Belgium
- Germany (3):
  - Universitätsklinikum Aachen, AÖR - Medizinische Fakultät der RWTH - Klinik für Urologie, Aachen
  - Universitätsklinikum "Carl Gustav Carus" Dresden - Klinik und Poliklinik für Urologie, Dresden
  - Klinikum Rechts der Isar - Urologische Klinik und Poliklinik, München

REFERENCES:
- [Derived] Wirth M, Heidenreich A, Gschwend JE, Gil T, Zastrow S, Laniado M, Gerloff J, Zuhlsdorf M, Mordenti G, Uhl W, Lannert H. A multicenter phase 1 study of EMD 525797 (DI17E6), a novel humanized monoclonal antibody targeting alphav integrins, in progressive castration-resistant prostate cancer with bone metastases after chemotherapy. Eur Urol. 2014 May;65(5):897-904. doi: 10.1016/j.eururo.2013.05.051. Epub 2013 Jun 6. PMID 23791392

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First/last subject (informed consent): 14 Oct 2008/21 May 2010. Last subject completed: 03 March 2011.
Groups:
- EMD 525797 250 mg: Subjects were administered with 250 milligram (mg) of EMD 525797 intravenously over 1 hour every 2 weeks for 6 weeks. Subjects who were clinically benefitted at the end of Week 6 continued at the same dose-level until disease progression, intolerance to treatment, withdrawal of consent or if the subject was no longer benefitted from the treatment as per Investigator's discretion.
- EMD 525797 500 mg: Subjects were administered with 500 mg of EMD 525797 intravenously over 1 hour every 2 weeks for 6 weeks. Subjects who were clinically benefitted at the end of Week 6 continued at the same dose-level until disease progression, intolerance to treatment, withdrawal of consent or if the subject was no longer benefitted from the treatment as per Investigator's discretion.
- EMD 525797 1000 mg: Subjects were administered with 1000 mg of EMD 525797 intravenously over 1 hour every 2 weeks for 6 weeks. Subjects who were clinically benefitted at the end of Week 6 continued at the same dose-level until disease progression, intolerance to treatment, withdrawal of consent or if the subject was no longer benefitted from the treatment as per Investigator's discretion.
- EMD 525797 1500 mg: Subjects were administered with 1500 mg of EMD 525797 intravenously over 1 hour every 2 weeks for 6 weeks. Subjects who were clinically benefitted at the end of Week 6 continued at the same dose-level until disease progression, intolerance to treatment, withdrawal of consent or if the subject was no longer benefitted from the treatment as per Investigator's discretion.
Period: Overall Study
Arm/Group | EMD 525797 250 mg | EMD 525797 500 mg | EMD 525797 1000 mg | EMD 525797 1500 mg
Started | 8 | 6 | 6 | 6
Completed | 8 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all subjects who received at least 1 dose of the study medication and had at least 1 follow-up safety measure.
Groups:
- Total: Total of all reporting groups
Arm/Group | EMD 525797 250 mg | EMD 525797 500 mg | EMD 525797 1000 mg | EMD 525797 1500 mg | Total
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.0 (6.0) | 63.0 (12.0) | 62.0 (12.0) | 66.0 (9.0) | 65.0 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 8 | 6 | 6 | 6 | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Dose Limiting Toxicity (DLT)
Description: DLT was defined using National Cancer Institute Common Toxicity Criteria for Adverse Events Version 3.0 as any Grade 3 or 4 hematological or non-hematological toxicity occurring at any dose level until the end of Week 6, and suspected to be reasonably related to the investigational product by the Investigator and/or Sponsor except for allergic/ hypersensitivity reactions and any Grade 3/4 out-of-range laboratory values without any clinical correlate, which were reversible within 7 days.
Time Frame: Baseline up to 6 weeks
Population: DLT analysis set: all subjects who experienced any DLT during first 6 weeks, regardless of number of doses of drug administered or who were considered completers (did not discontinue treatment for any reason other than DLT, were compliant, did not deviate in drug administration for more than +/-2 days due to any reason other than related toxicity).
Measure: Number; unit: subjects
Arm/Group | EMD 525797 250 mg | EMD 525797 500 mg | EMD 525797 1000 mg | EMD 525797 1500 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6
subjects | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Subjects With Treatment Emergent Adverse Events (TEAEs), Serious TEAEs and Related TEAEs
Description: An AE was defined as any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug or worsening of pre-existing medical condition, whether or not related to study drug. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. Treatment-emergent are events between first dose of study drug that were absent before treatment or that worsened relative to pre-treatment state. TEAEs include both Serious TEAEs and non-serious TEAEs.Treatment-related are events which had causal relationship to study drug as assessed by the Investigator and were suspected to be reasonably related to the study drug.
Time Frame: Baseline up to 534 days
Population: as for baseline characteristics
Measure: Number; unit: Subjects
Arm/Group | EMD 525797 250 mg | EMD 525797 500 mg | EMD 525797 1000 mg | EMD 525797 1500 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6
Subjects
  TEAEs | 8 | 6 | 6 | 6
  Serious TEAEs | 5 | 1 | 4 | 3
  Related TEAEs | 2 | 4 | 2 | 3

3. Primary Outcome: Observed Maximum Serum Concentration (Cmax) of EMD 525797 After First Infusion
Time Frame: pre-dose, end of infusion, 4, 8, 24, 48, 96, 168 and 336 hours post-infusion at Week 1
Population: Pharmacokinetic (PK) analysis set included all subjects who received at least first dose of the study drug according to the protocol and who provided sufficient data for a concentration time profile for EMD 525797.Here "Number of Participants analyzed" signifies those subjects who were evaluable for this outcome measure for each arm, respectively.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (mcg/mL)
Arm/Group | EMD 525797 250 mg | EMD 525797 500 mg | EMD 525797 1000 mg | EMD 525797 1500 mg
Number analyzed (Participants) | 8 | 5 | 6 | 6
microgram per milliliter (mcg/mL) | 52.9 (15.3) | 115.5 (20.1) | 298.0 (10.8) | 368.9 (26.7)

4. Primary Outcome: Observed Maximum Serum Concentration (Cmax) of EMD 525797 After Third Infusion
Time Frame: pre-dose, end of infusion, 4, 8, 24, 48, 96, 168 and 336 hours post-infusion at Week 5
Population: PK analysis set included all subjects who received at least the first dose of the study drug according to the protocol and who provided sufficient data for a concentration time profile for EMD 525797. Here "Number of Participants analyzed" signifies those subjects who were evaluable for this outcome measure for each arm, respectively.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | EMD 525797 250 mg | EMD 525797 500 mg | EMD 525797 1000 mg | EMD 525797 1500 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
mcg/mL | 55.7 (23.8) | 130.3 (17.0) | 371.8 (17.8) | 485.7 (25.0)

5. Primary Outcome: Area Under the Serum Concentration-time Curve From Time Zero to the Last Sampling Time (AUC0-t) After First Infusion
Description: Area under the serum concentration-time curve from time zero to the last sampling time at which the concentration is at or above lower limit of quantification (LLQ). AUC0-t was calculated according to the mixed log linear trapezoidal rule.
Time Frame: pre-dose, end of infusion, 4, 8, 24, 48, 96, 168 and 336 hours post-infusion at Week 1
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*mcg/mL
Arm/Group | EMD 525797 250 mg | EMD 525797 500 mg | EMD 525797 1000 mg | EMD 525797 1500 mg
Number analyzed (Participants) | 8 | 5 | 6 | 6
h*mcg/mL | 3583 (33) | 15609 (16) | 40080 (16) | 50891 (25)

6. Primary Outcome: Total Body Clearance of Drug From Serum (CL) After First Infusion
Description: Clearance of a drug was a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Total body clearance of drug from serum, calculated as CL = dose/AUC0-inf. Where AUC0-inf is area under the serum concentration time curve from time zero to infinity, calculated as AUC0 t + AUCextra. AUCextra represents an extrapolated value obtained by Clast/λz, where Clast is the calculated serum concentration at the last sampling time point at which the measured serum concentration is at or above lower limit of quantification (LLQ) and λz is elimination rate constant.
Time Frame: pre-dose, end of infusion, 4, 8, 24, 48, 96, 168 and 336 hours post-infusion at Week 1
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Groups:
- EMD 525797 1500 mg: Subjects were administered with 1000 mg of EMD 525797 intravenously over 1 hour every 2 weeks for 6 weeks. Subjects who were clinically benefitted at the end of Week 6 continued at the same dose-level until disease progression, intolerance to treatment, withdrawal of consent or if the subject was no longer benefitted from the treatment as per Investigator's discretion.
Arm/Group | EMD 525797 250 mg | EMD 525797 500 mg | EMD 525797 1000 mg | EMD 525797 1500 mg
Number analyzed (Participants) | 8 | 5 | 6 | 6
L/h | 0.060 (38.399) | 0.027 (25.827) | 0.019 (21.791) | 0.020 (28.933)

7. Primary Outcome: Apparent Volume of Distribution During Terminal Phase (Vz) of EMD 525797 After First Infusion
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired serum concentration of a drug. Apparent volume of distribution during the terminal phase, calculated as = Dose/(AUC0-inf *λz) after first infusion. Where 'λz' is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve. Where AUC0-inf is area under the serum concentration time curve from time zero to infinity, calculated as AUC0 t + AUCextra. AUCextra represents an extrapolated value obtained by Clast/λz, where Clast is the calculated serum concentration at the last sampling time point at which the measured serum concentration is at or above lower limit of quantification (LLQ) and λz is elimination rate constant.
Time Frame: pre-dose, end of infusion, 4, 8, 24, 48, 96, 168 and 336 hours post-infusion at Week 1
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | EMD 525797 250 mg | EMD 525797 500 mg | EMD 525797 1000 mg | EMD 525797 1500 mg
Number analyzed (Participants) | 8 | 5 | 6 | 6
Liters | 5.06 (17.49) | 4.64 (7.83) | 4.35 (34.54) | 6.16 (24.13)

8. Primary Outcome: Trough Serum Concentration (Ctrough) Of EMD 525797 at Week 1
Description: Ctrough is the concentration prior to study drug administration.
Time Frame: pre-dose at Week 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | EMD 525797 250 mg | EMD 525797 500 mg | EMD 525797 1000 mg | EMD 525797 1500 mg
Number analyzed (Participants) | 7 | 5 | 6 | 6
mcg/mL | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)

9. Primary Outcome: Trough Serum Concentration (Ctrough) Of EMD 525797 at Week 3
Description: Ctrough is the concentration prior to study drug administration.
Time Frame: pre-dose at Week 3
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | EMD 525797 250 mg | EMD 525797 500 mg | EMD 525797 1000 mg | EMD 525797 1500 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
mcg/mL | 0.43 (1.05) | 15.17 (6.97) | 51.16 (23.46) | 81.22 (26.72)

10. Primary Outcome: Trough Serum Concentration (Ctrough) Of EMD 525797 at Week 5
Description: Ctrough is the concentration prior to study drug administration.
Time Frame: pre-dose at Week 5
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | EMD 525797 250 mg | EMD 525797 500 mg | EMD 525797 1000 mg | EMD 525797 1500 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
mcg/mL | 2.70 (4.05) | 27.97 (12.33) | 105.77 (25.22) | 150.74 (47.37)

11. Secondary Outcome: Time to Reach Observed Serum Concentration (Tmax) After First Infusion
Time Frame: pre-dose, end of infusion, 4, 8, 24, 48, 96, 168 and 336 hours post-infusion at Week 1
Population: as for outcome 4
Measure: Median (Full Range); unit: hours
Arm/Group | EMD 525797 250 mg | EMD 525797 500 mg | EMD 525797 1000 mg | EMD 525797 1500 mg
Number analyzed (Participants) | 8 | 5 | 6 | 6
hours | 1.0 [1.0 to 5.0] | 8 [1 to 24] | 2.0 [1.0 to 4.0] | 2.0 [1.0 to 5.0]

12. Secondary Outcome: Time to Reach Observed Serum Concentration (Tmax) After Third Infusion
Time Frame: pre-dose, end of infusion, 4, 8, 24, 48, 96, 168 and 336 hours post-infusion at Week 5
Population: as for outcome 4
Measure: Median (Full Range); unit: hours
Arm/Group | EMD 525797 250 mg | EMD 525797 500 mg | EMD 525797 1000 mg | EMD 525797 1500 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
hours | 1 [1 to 5] | 3 [1 to 5] | 1 [1 to 4] | 1 [1 to 8]

13. Secondary Outcome: Number of Subjects With Positive Anti-EMD 525797 Antibodies
Time Frame: Week 1, 3, 5, 8, 9
Population: as for baseline characteristics
Measure: Number; unit: Subjects
Arm/Group | EMD 525797 250 mg | EMD 525797 500 mg | EMD 525797 1000 mg | EMD 525797 1500 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6
Subjects
  Week 1 | 0 | 0 | 0 | 0
  Week 3 | 4 | 0 | 0 | 0
  Week 5 | 1 | 0 | 0 | 0
  Week 8 | 1 | 0 | 0 | 0
  Week 9 | 1 | 0 | 0 | 0

14. Secondary Outcome: Serum Levels of Interleukin 6 (IL-6) and Interleukin 8 (IL-8)
Time Frame: Week 1 up to a maximum of 56 days
Population: As per change in planned analysis, it was decided that that the biomarker analysis were not significantly associated with compound administration and thus the data was not collected for this outcome.
Groups:
- EMD 525797 250 mg: Subjects were administered with 250 milligram (mg) mg of EMD 525797 intravenously over 1 hour every 2 weeks for 6 weeks. Subjects who will be clinically benefitted at the end of Week 6 will continue at the same dose-level until disease progression, intolerance to treatment, withdrawal of consent or if the subject was no longer benefitted from the treatment as per Investigator's discretion.
- EMD 525797 500 mg: Subjects were administered with 500 mg of EMD 525797 intravenously over 1 hour every 2 weeks for 6 weeks. Subjects who will be clinically benefitted at the end of Week 6 will continue at the same dose-level until disease progression, intolerance to treatment, withdrawal of consent or if the subject was no longer benefitted from the treatment as per Investigator's discretion.
- EMD 525797 1000 mg: Subjects were administered with 1000 mg of EMD 525797 intravenously over 1 hour every 2 weeks for 6 weeks. Subjects who will be clinically benefitted at the end of Week 6 will continue at the same dose-level until disease progression, intolerance to treatment, withdrawal of consent or if the subject was no longer benefitted from the treatment as per Investigator's discretion.
- EMD 525797 1500 mg: Subjects were administered with 1500 mg of EMD 525797 intravenously over 1 hour every 2 weeks for 6 weeks. Subjects who will be clinically benefitted at the end of Week 6 will continue at the same dose-level until disease progression, intolerance to treatment, withdrawal of consent or if the subject was no longer benefitted from the treatment as per Investigator's discretion.
Arm/Group | EMD 525797 250 mg | EMD 525797 500 mg | EMD 525797 1000 mg | EMD 525797 1500 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

15. Secondary Outcome: C-Reactive Protein Levels
Time Frame: Week 1 up to a maximum of 56 days
Population: as for outcome 14
Groups:
- EMD 525797 1500 mg: Subjects were administered with 1000 mg of EMD 525797 intravenously over 1 hour every 2 weeks for 6 weeks. Subjects who will be clinically benefitted at the end of Week 6 will continue at the same dose-level until disease progression, intolerance to treatment, withdrawal of consent or if the subject was no longer benefitted from the treatment as per Investigator's discretion.
Arm/Group | EMD 525797 250 mg | EMD 525797 500 mg | EMD 525797 1000 mg | EMD 525797 1500 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

16. Secondary Outcome: Apparent Terminal Half-life (t1/2) of EMD 525797 After First Infusion
Description: Terminal half-life is the time measured for the concentration to decrease by one half. Terminal half-life is calculated by dividing the natural logarithm to the base e (Log e) multiplied by (*) 2/ λz, where 'λz' is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: pre-dose, end of infusion, 4, 8, 24, 48, 96, 168 and 336 hours post-infusion at Week 1
Population: as for outcome 4
Measure: Median (Full Range); unit: hours
Arm/Group | EMD 525797 250 mg | EMD 525797 500 mg | EMD 525797 1000 mg | EMD 525797 1500 mg
Number analyzed (Participants) | 8 | 5 | 6 | 6
hours | 60.3 [31.3 to 88.7] | 109.5 [92.0 to 186.8] | 184.5 [66.3 to 233.1] | 222.1 [174.7 to 257.6]

17. Secondary Outcome: Elimination Rate Constant (λz) of EMD 525797 After First Infusion
Description: Elimination rate constant obtained from linear regression of the terminal phase of the log transformed concentration-time data.
Time Frame: pre-dose, end of infusion, 4, 8, 24, 48, 96, 168 and 336 hours post-infusion at Week 1
Population: PK analysis set included all subjects who received at least first dose of the study drug according to the protocol and who provided sufficient data for a concentration time profile for EMD 525797. Here "Number of Participants analyzed" signifies those subjects who were evaluable for this outcome measure for each arm, respectively.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/h
Arm/Group | EMD 525797 250 mg | EMD 525797 500 mg | EMD 525797 1000 mg | EMD 525797 1500 mg
Number analyzed (Participants) | 8 | 5 | 6 | 6
1/h | 0.0119 (34.2179) | 0.0059 (28.8297) | 0.0043 (47.9226) | 0.0032 (16.6282)

18. Secondary Outcome: Observed Minimum Serum Concentration (Cmin) of EMD 525797 After Third Infusion
Description: Observed minimum serum concentration determined directly from the serum concentration-time profile of each subject.
Time Frame: pre-dose, end of infusion, 4, 8, 24, 48, 96, 168 and 336 hours post-infusion at Week 5
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | EMD 525797 250 mg | EMD 525797 500 mg | EMD 525797 1000 mg | EMD 525797 1500 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
mcg/mL | 2.7 (4.1) | 28.0 (12.3) | 102.8 (28.2) | 150.7 (47.4)

19. Secondary Outcome: Average Serum Concentration at Steady State (Cav) of EMD 525797 After Third Infusion
Description: The average serum concentration at steady state, calculated as Cav = AUCtau/tau, where tau is the dosing interval (336 hours).
Time Frame: pre-dose, end of infusion, 4, 8, 24, 48, 96, 168, 336 hours post third infusion at Week 5
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | EMD 525797 250 mg | EMD 525797 500 mg | EMD 525797 1000 mg | EMD 525797 1500 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
mcg/mL | 16.4 (59.6) | 57.1 (41.9) | 187.2 (28.2) | 178.5 (41.3)

20. Secondary Outcome: Area Under the Serum Concentration-time Curve Within One Complete Dosing Interval (AUCtau) of EMD 525797 After First Infusion
Description: Area under the concentration-time curve from time zero up to time Tau, where Tau is the dosing interval (168 hours).
Time Frame: pre-dose, end of infusion, 4, 8, 24, 48, 96 and 168 hours post-infusion at Week 1
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*mcg/mL
Arm/Group | EMD 525797 250 mg | EMD 525797 500 mg | EMD 525797 1000 mg | EMD 525797 1500 mg
Number analyzed (Participants) | 6 | 5 | 6 | 6
h*mcg/mL | 4398 (33) | 15609 (16) | 40080 (16) | 50553 (24)

21. Secondary Outcome: Area Under the Serum Concentration-time Curve Within One Complete Dosing Interval (AUCtau) of EMD 525797 After Third Infusion
Description: Area under the concentration-time curve from time zero up to time Tau, where Tau is the dosing interval (336 hours).
Time Frame: pre-dose, end of infusion, 4, 8, 24, 48, 96,168, 336 hours post third infusion at Week 5
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*mcg/mL
Arm/Group | EMD 525797 250 mg | EMD 525797 500 mg | EMD 525797 1000 mg | EMD 525797 1500 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
h*mcg/mL | 6028 (50) | 20306 (35) | 67160 (19) | 85401 (25)

22. Secondary Outcome: Area Under the Serum Concentration-time Curve From Time Zero to Infinity (AUC0-inf) of EMD 525797 After First Infusion
Description: Area under the serum concentration time curve from time zero to infinity, calculated as AUC0 t + AUCextra. AUCextra represents an extrapolated value obtained by Clast/λz, where Clast is the calculated serum concentration at the last sampling time point at which the measured serum concentration is at or above LLQ and λz is elimination rate constant.
Time Frame: pre-dose, end of infusion, 4, 8, 24, 48, 96, 168 and 336 hours post-infusion at Week 1
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*mcg/mL
Arm/Group | EMD 525797 250 mg | EMD 525797 500 mg | EMD 525797 1000 mg | EMD 525797 1500 mg
Number analyzed (Participants) | 8 | 5 | 6 | 6
h*mcg/mL | 4152 (38) | 18317 (26) | 53580 (22) | 75408 (29)

23. Secondary Outcome: Peak Trough Fluctuation Over One Dosing Interval at Steady State (%PTF) of EMD 525797 After Third Infusion
Description: The peak trough fluctuation over one dosing interval at steady state, calculated as PTF (%) = ( [ Cmax - Cmin ] / Cav )*100
Time Frame: pre-dose, end of infusion, 4, 8, 24, 48, 96, 168 and 336 hours post-infusion at Week 5
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of fluctuation
Arm/Group | EMD 525797 250 mg | EMD 525797 500 mg | EMD 525797 1000 mg | EMD 525797 1500 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
percentage of fluctuation | 326 (39) | 179 (43) | 145 (18) | 190 (32)

24. Secondary Outcome: Mean Residence Time of Drug in the Body (MRT) of EMD 525797 After First Infusion
Description: Mean residence time of drug in the body calculated as: AUMC0-inf / AUC0-inf, where AUMC0-inf is the area under the first moment curve from time zero to infinity. Where AUC0-inf is area under the serum concentration time curve from time zero to infinity, calculated as AUC0 t + AUCextra. AUCextra represents an extrapolated value obtained by Clast/λz, where Clast is the calculated serum concentration at the last sampling time point at which the measured serum concentration is at or above lower limit of quantification (LLQ) and λz is elimination rate constant.
Time Frame: pre-dose, end of infusion, 4, 8, 24, 48, 96, 168 and 336 hours post-infusion at Week 1
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | EMD 525797 250 mg | EMD 525797 500 mg | EMD 525797 1000 mg | EMD 525797 1500 mg
Number analyzed (Participants) | 8 | 5 | 6 | 6
hours | 87.2 (33.3) | 171.0 (26.6) | 230.5 (41.3) | 299.9 (16.2)

25. Secondary Outcome: Apparent Volume of Distribution at Steady State (Vss) of EMD 525797 After Third Infusion
Description: Apparent volume of distribution at steady-state was reported. Apparent volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired serum concentration of a drug.
Time Frame: pre-dose, end of infusion, 4, 8, 24, 48, 96, 168 and 336 hours post-infusion at Week 5
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | EMD 525797 250 mg | EMD 525797 500 mg | EMD 525797 1000 mg | EMD 525797 1500 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
Liters | 4.63 (24.42) | 4.35 (3.79) | 3.35 (10.55) | 4.32 (29.04)

26. Secondary Outcome: Accumulation Ratio Of Cmax (R_Cmax)
Description: Accumulation ratio for Cmax was calculated as Cmax, after third dose/Cmax, after first dose.
Time Frame: pre-dose, end of infusion, 4, 8, 24, 48, 96, 168 and 336 hours post-infusion at Week 1 and Week 5
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | EMD 525797 250 mg | EMD 525797 500 mg | EMD 525797 1000 mg | EMD 525797 1500 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
ratio | 1.10 (15.13) | 1.19 (18.25) | 1.25 (9.84) | 1.32 (14.59)

27. Secondary Outcome: Accumulation Ratio of AUC (R_AUC)
Description: Accumulation ratio for AUC, calculated as area under the serum concentration-time curve within one complete dosing interval at third dose divided by area under the serum concentration-time curve within one complete dosing interval at first dose.
Time Frame: pre-dose, end of infusion, 4, 8, 24, 48, 96,168 hours post-infusion at Week 1 and pre-dose, end of infusion, 4, 8, 24, 48, 96, 168, 336 hours post third infusion at Week 5
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | EMD 525797 250 mg | EMD 525797 500 mg | EMD 525797 1000 mg | EMD 525797 1500 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
ratio | 1.37 (29.43) | 1.32 (28.35) | 1.68 (18.91) | 1.69 (10.31)

28. Secondary Outcome: Number of Subjects With Best Overall Response (BOR)
Description: Number of subjects with BOR in each category (complete response [CR], partial response [PR], stable disease [SD], progressive disease [PD]) according to Response Evaluation Criteria in Solid Tumors (RECIST Version 1.0) was reported. CR: defined as disappearance of all target and all non-target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: defined as at least a 30% decrease in sum of longest diameter of target lesions, taking as reference the baseline sum of longest diameter. PD:defined as at least a 20% increase in sum of longest diameter of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study) or unequivocal progression of existing non-target lesions. SD: defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of longest diameter while on study.
Time Frame: Week 6, Week 19, Overall (Baseline Up to 394 days)
Population: Efficacy analysis set included all subjects who received at least 1 dose of the study drug.
Measure: Number; unit: subjects
Arm/Group | EMD 525797 250 mg | EMD 525797 500 mg | EMD 525797 1000 mg | EMD 525797 1500 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6
subjects
  Week 6: CR | 0 | 0 | 0 | 0
  Week 6: PR | 0 | 0 | 0 | 0
  Week 6: SD | 4 | 5 | 4 | 5
  Week 6: PD | 4 | 1 | 2 | 1
  Week 19: CR | 0 | 0 | 0 | 0
  Week 19: PR | 0 | 1 | 0 | 0
  Week 19: SD | 4 | 4 | 4 | 5
  Week 19: PD | 4 | 1 | 2 | 1
  Overall: CR | 0 | 0 | 0 | 0
  Overall: PR | 0 | 1 | 0 | 0
  Overall: SD | 4 | 4 | 4 | 5
  Overall: PD | 4 | 1 | 2 | 1

29. Secondary Outcome: Progression-free Survival (PFS) as Per Prostate Cancer Clinical Trials Working Group 1 (PCWG1) and Prostate Cancer Clinical Trials Working Group 2 (PCWG2) Criteria
Description: PFS PCWG1 criteria: time from the day treatment is initiated up to progression (for subject's whose prostate specific antigen [PSA] level did not decrease after baseline, progression defined as 50% PSA increase relative to baseline; for subject's whose PSA decreased after baseline, progression defined as 50% PSA increase relative to nadir [smallest PSA value post-baseline]. Progression was confirmed if progression criterion was met in next 2 assessments as well.) PFS PCWG2 criteria: time from study entry to disease progression or death. Progression was defined as first appearance of progression according to PSA (for subject's whose PSA decreased after baseline, progression was defined as 25% PSA increase relative to nadir. Progression was confirmed if another assessment measured at least 3 weeks later met the criterion as well; for subject's whose PSA did not decrease after baseline, progression was defined as 25% PSA increase relative to baseline assessed 12 weeks after baseline).
Time Frame: Baseline up to 394 days
Population: Efficacy analysis set included all subjects who received at least 1 dose of the study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | EMD 525797 250 mg | EMD 525797 500 mg | EMD 525797 1000 mg | EMD 525797 1500 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6
months
  PCWG1 | NA [1.4 to NA] — Median and corresponding upper limit of confidence interval could not be estimated by Kaplan-Meier method due to limited number of events. | 1.0 [1.0 to 1.4] | 2.3 [1.4 to 2.3] | 7.5 [2.6 to 7.5]
  PCWG2 | 3.0 [1.7 to 3.7] | 3.4 [1.8 to NA] — Upper limit of confidence interval could not be estimated by Kaplan-Meier method due to limited number of events. | 3.9 [2.0 to 4.7] | 3.4 [2.3 to 5.4]

30. Secondary Outcome: Time to Progression (TTP)
Description: TTP was calculated as the time between the date of imaging for the earliest visit where progressive disease was detected and the first dose date plus 1 day. Participants without event are censored on the date of last tumor assessment.
Time Frame: Baseline up to disease progression up to a maximum of 13.1 months
Population: Efficacy analysis set included all subjects who received at least 1 dose of the study drug. Here "Number of Participants" analyzed signifies those subjects who were evaluable for this outcome measure.
Measure: Number; unit: months
Arm/Group | EMD 525797 250 mg | EMD 525797 500 mg | EMD 525797 1000 mg | EMD 525797 1500 mg
Number analyzed (Participants) | 3 | 2 | 2 | 2
months
  Subject 1 | 1.18 | 4.17 | 1.28 | 2.83
  Subject 2 | 3.02 | 1.18 | 1.25 | 1.18
  Subject 3 | 1.48 | NA — there were only 2 subjects who reported an event for the specified arm | NA — there were only 2 subjects who reported an event for the specified arm | NA — there were only 2 subjects who reported an event for the specified arm

31. Secondary Outcome: Number of Subjects With Eastern Cooperative Oncology Group (ECOG) Performance: Baseline Score vs. Worst Post-baseline Score
Description: ECOG performance status measured to assess subject's performance status on a scale of 0 to 4, where 0=Fully active, able to carry on all pre-disease activities without restriction; 1=Restricted in physically strenuous activity, ambulatory and able to carry out light or sedentary work; 2=Ambulatory (>50% of waking hours), capable of all self-care, unable to carry out any work activities; 3=Capable of only limited self-care, confined to bed/chair >50% of waking hours; 4=Completely disabled, cannot carry on any self-care, totally confined to bed/chair. ECOG performance status was reported in terms of number of subjects with Baseline value vs. worst post-baseline value (i.e. highest score) combination.
Time Frame: Baseline up to 394 days
Population: as for baseline characteristics
Measure: Number; unit: subjects
Arm/Group | EMD 525797 250 mg | EMD 525797 500 mg | EMD 525797 1000 mg | EMD 525797 1500 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6
subjects
  Baseline score 0, worst post-baseline score 0 | 2 | 3 | 2 | 1
  Baseline score 0, worst post-baseline score 1 | 1 | 0 | 1 | 0
  Baseline score 0, worst post-baseline score 2 | 0 | 0 | 0 | 1
  Baseline score 0, worst post-baseline score 3 | 0 | 0 | 0 | 1
  Baseline score 0, worst post-baseline score 4 | 0 | 0 | 0 | 0
  Baseline score 1, worst post-baseline score 0 | 1 | 0 | 0 | 0
  Baseline score 1, worst post-baseline score 1 | 2 | 3 | 2 | 1
  Baseline score 1, worst post-baseline score 2 | 1 | 0 | 0 | 1
  Baseline score 1, worst post-baseline score 3 | 1 | 0 | 0 | 0
  Baseline score 1, worst post-baseline score 4 | 0 | 0 | 0 | 0
  Baseline score 2, worst post-baseline score 0 | 0 | 0 | 0 | 0
  Baseline score 2, worst post-baseline score 1 | 0 | 0 | 0 | 1
  Baseline score 2, worst post-baseline score 2 | 0 | 0 | 0 | 0
  Baseline score 2, worst post-baseline score 3 | 0 | 0 | 1 | 0
  Baseline score 2, worst post-baseline score 4 | 0 | 0 | 0 | 0
  Baseline score 3, worst post-baseline score 0 | 0 | 0 | 0 | 0
  Baseline score 3, worst post-baseline score 1 | 0 | 0 | 0 | 0
  Baseline score 3, worst post-baseline score 2 | 0 | 0 | 0 | 0
  Baseline score 3, worst post-baseline score 3 | 0 | 0 | 0 | 0
  Baseline score 3, worst post-baseline score 4 | 0 | 0 | 0 | 0
  Baseline score 4, worst post-baseline score 0 | 0 | 0 | 0 | 0
  Baseline score 4, worst post-baseline score 1 | 0 | 0 | 0 | 0
  Baseline score 4, worst post-baseline score 2 | 0 | 0 | 0 | 0
  Baseline score 4, worst post-baseline score 3 | 0 | 0 | 0 | 0
  Baseline score 4, worst post-baseline score 4 | 0 | 0 | 0 | 0

32. Secondary Outcome: Number of Subjects With Eastern Cooperative Oncology Group (ECOG) Performance: Baseline Score vs. Best Post-baseline Score
Description: ECOG performance status measured to assess subject's performance status on a scale of 0 to 4, where 0=Fully active, able to carry on all pre-disease activities without restriction; 1=Restricted in physically strenuous activity, ambulatory and able to carry out light or sedentary work; 2=Ambulatory (>50% of waking hours), capable of all self-care, unable to carry out any work activities; 3=Capable of only limited self-care, confined to bed/chair >50% of waking hours; 4=Completely disabled, cannot carry on any self-care, totally confined to bed/chair. ECOG performance status was reported in terms of number of subjects with Baseline value vs. best post-baseline value (i.e. lowest score) combination.
Time Frame: Baseline up to 394 days
Population: as for baseline characteristics
Measure: Number; unit: subjects
Arm/Group | EMD 525797 250 mg | EMD 525797 500 mg | EMD 525797 1000 mg | EMD 525797 1500 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6
subjects
  Baseline score 0, best post-baseline score 0 | 3 | 3 | 3 | 3
  Baseline score 0, best post-baseline score 1 | 0 | 0 | 0 | 0
  Baseline score 0, best post-baseline score 2 | 0 | 0 | 0 | 0
  Baseline score 0, best post-baseline score 3 | 0 | 0 | 0 | 0
  Baseline score 0, best post-baseline score 4 | 0 | 0 | 0 | 0
  Baseline score 1, best post-baseline score 0 | 3 | 2 | 0 | 1
  Baseline score 1, best post-baseline score 1 | 1 | 1 | 2 | 1
  Baseline score 1, best post-baseline score 2 | 1 | 0 | 0 | 0
  Baseline score 1, best post-baseline score 3 | 0 | 0 | 0 | 0
  Baseline score 1, best post-baseline score 4 | 0 | 0 | 0 | 0
  Baseline score 2, best post-baseline score 0 | 0 | 0 | 0 | 1
  Baseline score 2, best post-baseline score 1 | 0 | 0 | 0 | 0
  Baseline score 2, best post-baseline score 2 | 0 | 0 | 1 | 0
  Baseline score 2, best post-baseline score 3 | 0 | 0 | 0 | 0
  Baseline score 2, best post-baseline score 4 | 0 | 0 | 0 | 0
  Baseline score 3, best post-baseline score 0 | 0 | 0 | 0 | 0
  Baseline score 3, best post-baseline score 1 | 0 | 0 | 0 | 0
  Baseline score 3, best post-baseline score 2 | 0 | 0 | 0 | 0
  Baseline score 3, best post-baseline score 3 | 0 | 0 | 0 | 0
  Baseline score 3, best post-baseline score 4 | 0 | 0 | 0 | 0
  Baseline score 4, best post-baseline score 0 | 0 | 0 | 0 | 0
  Baseline score 4, best post-baseline score 1 | 0 | 0 | 0 | 0
  Baseline score 4, best post-baseline score 2 | 0 | 0 | 0 | 0
  Baseline score 4, best post-baseline score 3 | 0 | 0 | 0 | 0
  Baseline score 4, best post-baseline score 4 | 0 | 0 | 0 | 0

33. Secondary Outcome: Total Pain Score Using Brief Pain Inventory-Short Form (BPI-sf)
Description: BPI-sf is an 11-item self-report questionnaire that is designed to assess the severity and impact of pain on daily functions. BPI-sf has 4 questions that assess pain intensity (worst, least, average, right now) and 7 questions that assess impact of pain on daily functions (general activity, mood, walking ability, normal work, relations with other people, sleep, enjoyment of life). Each question is answered on a scale ranging from 0 to 10;'0=No pain and 10=Pain as bad as you can imagine'.Total score is reported as average of individual questions ranges from 0 to 10, with lower scores being indicative of less pain or pain interference.Data was not available for "EMD 525797 250 mg" arm for FUP Weeks 15, 19, 23, 27, 31, 35, 39, 43, 47, 51, 55, 59, 63, 67, 71, 75 and "EMD 525797 1000 mg" arm for FUP Weeks 47, 51, 55, 59, 63, 67, 71 and "EMD 525797 1500 mg arm" for FUP Weeks 35, 39, 43, 47, 51, 55, 59, 63, 67, 71, 75 respectively as no subjects were evaluable at the specified FUP visits.
Time Frame: Screening; Baseline; Week 3, 5, 7; Follow-up (FUP) Week 11, 15, 19, 23, 27, 31, 35, 39, 43, 47, 51, 55, 59, 63, 67, 71, 75; End of treatment (EOT; maximum up to 380 days) and EOS (maximum up to 394 days)
Population: Efficacy analysis set included all subjects who received at least 1 dose of the study drug. Here "n" signifies those subjects who were evaluable for this outciome measure at the specified time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EMD 525797 250 mg | EMD 525797 500 mg | EMD 525797 1000 mg | EMD 525797 1500 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6
score on a scale
  Screening | 2.32 (2.34) | 1.95 (1.29) | 1.95 (2.15) | 2.52 (3.13)
  Baseline | 1.73 (1.57) | 1.64 (1.80) | 1.71 (1.88) | 2.62 (3.84)
  Week 3: number analyzed (Participants) | 7 | 6 | 6 | 6
  Week 3 | 1.98 (1.98) | 2.57 (1.79) | 2.24 (1.82) | 1.87 (2.48)
  Week 5: number analyzed (Participants) | 6 | 6 | 6 | 6
  Week 5 | 2.21 (2.27) | 2.29 (2.32) | 2.36 (2.73) | 1.86 (2.43)
  Week 7: number analyzed (Participants) | 6 | 6 | 5 | 6
  Week 7 | 2.38 (2.92) | 2.17 (1.62) | 2.31 (3.06) | 1.86 (1.92)
  FUP Week 11: number analyzed (Participants) | 1 | 4 | 3 | 4
  FUP Week 11 | 0.00 (NA) — Standard deviation could not be calculated as there was only 1 subjects analyzed at the specified FUP visit. | 3.00 (0.87) | 1.33 (1.73) | 4.75 (3.17)
  FUP Week 15: number analyzed (Participants) | 0 | 4 | 2 | 2
  FUP Week 15 |  | 2.68 (0.65) | 2.21 (2.73) | 3.43 (4.85)
  FUP Week 19: number analyzed (Participants) | 0 | 3 | 1 | 2
  FUP Week 19 |  | 3.33 (1.95) | 0.57 (NA) — Standard deviation could not be calculated as there was only 1 subjects analyzed at the specified FUP visit. | 3.29 (3.43)
  FUP Week 23: number analyzed (Participants) | 0 | 2 | 1 | 2
  FUP Week 23 |  | 2.36 (0.51) | 1.00 (NA) — Standard deviation could not be calculated as there was only 1 subjects analyzed at the specified FUP visit. | 2.57 (3.64)
  FUP Week 27: number analyzed (Participants) | 0 | 2 | 1 | 1
  FUP Week 27 |  | 1.57 (0.40) | 1.00 (NA) — Standard deviation could not be calculated as there was only 1 subjects analyzed at the specified FUP visit. | 1.57 (NA) — Standard deviation could not be calculated as there was only 1 subjects analyzed at the specified FUP visit.
  FUP Week 31: number analyzed (Participants) | 0 | 2 | 1 | 1
  FUP Week 31 |  | 1.93 (0.51) | 1.00 (NA) — Standard deviation could not be calculated as there was only 1 subjects analyzed at the specified FUP visit. | 0.00 (NA) — Standard deviation could not be calculated as there was only 1 subjects analyzed at the specified FUP visit.
  FUP Week 35: number analyzed (Participants) | 0 | 2 | 1 | 0
  FUP Week 35 |  | 2.29 (0.20) | 1.14 (NA) — Standard deviation could not be calculated as there was only 1 subjects analyzed at the specified FUP visit. |
  FUP Week 39: number analyzed (Participants) | 0 | 2 | 1 | 0
  FUP Week 39 |  | 2.50 (0.51) | 1.43 (NA) — Standard deviation could not be calculated as there was only 1 subjects analyzed at the specified FUP visit. |
  FUP Week 43: number analyzed (Participants) | 0 | 2 | 1 | 0
  FUP Week 43 |  | 5.00 (3.03) | 1.86 (NA) — Standard deviation could not be calculated as there was only 1 subjects analyzed at the specified FUP visit. |
  FUP Week 47: number analyzed (Participants) | 0 | 1 | 0 | 0
  FUP Week 47 |  | 2.00 (NA) — Standard deviation could not be calculated as there was only 1 subjects analyzed at the specified FUP visit. |  |
  FUP Week 51: number analyzed (Participants) | 0 | 1 | 0 | 0
  FUP Week 51 |  | 3.00 (NA) — Standard deviation could not be calculated as there was only 1 subjects analyzed at the specified FUP visit. |  |
  FUP Week 55: number analyzed (Participants) | 0 | 1 | 0 | 0
  FUP Week 55 |  | 3.00 (NA) — Standard deviation could not be calculated as there was only 1 subjects analyzed at the specified FUP visit. |  |
  FUP Week 59: number analyzed (Participants) | 0 | 1 | 0 | 0
  FUP Week 59 |  | 2.71 (NA) — Standard deviation could not be calculated as there was only 1 subjects analyzed at the specified FUP visit. |  |
  FUP Week 63: number analyzed (Participants) | 0 | 1 | 0 | 0
  FUP Week 63 |  | 2.57 (NA) — Standard deviation could not be calculated as there was only 1 subjects analyzed at the specified FUP visit. |  |
  FUP Week 67: number analyzed (Participants) | 0 | 1 | 0 | 0
  FUP Week 67 |  | 2.43 (NA) — Standard deviation could not be calculated as there was only 1 subjects analyzed at the specified FUP visit. |  |
  FUP Week 71: number analyzed (Participants) | 0 | 1 | 0 | 0
  FUP Week 71 |  | 2.29 (NA) — Standard deviation could not be calculated as there was only 1 subjects analyzed at the specified FUP visit. |  |
  FUP Week 75: number analyzed (Participants) | 0 | 1 | 0 | 0
  FUP Week 75 |  | 2.43 (NA) — Standard deviation could not be calculated as there was only 1 subjects analyzed at the specified FUP visit. |  |
  EOT: number analyzed (Participants) | 3 | 2 | 2 | 2
  EOT | 2.19 (2.76) | 3.36 (3.74) | 1.50 (0.10) | 3.41 (1.24)
  EOS: number analyzed (Participants) | 3 | 5 | 4 | 4
  EOS | 1.86 (3.22) | 3.63 (3.70) | 2.82 (2.22) | 2.71 (2.12)

34. Secondary Outcome: Maximum Percent Change From Baseline in Prostate Specific Antigen (PSA) Level
Description: Maximum percent change from Baseline in PSA Level during the study was reported.
Time Frame: Baseline up to 394 days
Population: Efficacy analysis set included all subjects who received at least 1 dose of the study drug.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | EMD 525797 250 mg | EMD 525797 500 mg | EMD 525797 1000 mg | EMD 525797 1500 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6
percent change | 138.41 (234.40) | 580.32 (1083.12) | 120.76 (108.18) | 120.41 (159.14)

35. Secondary Outcome: Minimum Percent Change From Baseline in PSA Level
Description: Minimum percent change from Baseline in PSA Level during the study was reported.
Time Frame: Baseline up to 394 days
Population: Efficacy analysis set included all subjects who received at least 1 dose of the study drug.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | EMD 525797 250 mg | EMD 525797 500 mg | EMD 525797 1000 mg | EMD 525797 1500 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6
percent change | 8.69 (21.91) | -9.88 (63.59) | 17.94 (9.16) | -7.72 (34.74)

ADVERSE EVENTS:
Time Frame: Baseline up to 394 days
Arm/Group | EMD 525797 250 mg | EMD 525797 500 mg | EMD 525797 1000 mg | EMD 525797 1500 mg
Serious Adverse Events (participants affected / at risk) | 5/8 | 1/6 | 4/6 | 3/6
Other Adverse Events (participants affected / at risk) | 8/8 | 6/6 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EMD 525797 250 mg (N=8) | EMD 525797 500 mg (N=6) | EMD 525797 1000 mg (N=6) | EMD 525797 1500 mg (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Anaemia Of Malignant Disease (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Euthanasia (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Bile Duct Stone (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 1 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain In Jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Metastases To Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Paraplegia (Nervous system disorders) | 1 | 0 | 0 | 0
Ureteric Obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 0
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EMD 525797 250 mg (N=8) | EMD 525797 500 mg (N=6) | EMD 525797 1000 mg (N=6) | EMD 525797 1500 mg (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Vision Blurred (Eye disorders) | 0 | 1 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Abdominal Tenderness (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Dry Mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hypoaesthesia Oral (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Swollen Tongue (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 2 | 2
General Physical Health Deterioration (General disorders) | 1 | 0 | 1 | 1
Infusion Site Extravasation (General disorders) | 0 | 0 | 0 | 1
Mucosal Inflammation (General disorders) | 0 | 0 | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 0 | 1 | 0 | 0
Oedema Peripheral (General disorders) | 2 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Bile Duct Stone (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1
Cystitis Escherichia (Infections and infestations) | 0 | 0 | 1 | 0
Fungal Infection (Infections and infestations) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 1
Rhinitis (Infections and infestations) | 1 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 2 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Joint Sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 1 | 0 | 0
Blood Creatinine Increased (Investigations) | 1 | 0 | 0 | 0
Blood Pressure Increased (Investigations) | 0 | 1 | 0 | 0
Gamma-Glutamyltransferase Increased (Investigations) | 1 | 1 | 0 | 0
Haemoglobin Decreased (Investigations) | 0 | 1 | 0 | 0
Weight Decreased (Investigations) | 0 | 0 | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 1
Pain In Jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0
Bladder Pain (Renal and urinary disorders) | 0 | 1 | 0 | 0
Micturition Disorder (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 1 | 0 | 0
Balanitis (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 1 | 0
Peripheral Coldness (Vascular disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No